CLINICAL TRIAL: NCT01726062
Title: Motivational Incentives to Reduce Secondhand Smoke in NICU Infants' Homes (The Baby's Breath II Project)
Brief Title: Motivational Incentives to Reduce Secondhand Smoke in NICU Infants' Homes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Memorial Hermann Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Angela Stotts, Associate Professor - Family Medicine, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-11-0641; 1R01HL107404-01A1 (NIH)
Record Dates: First submitted 2012-11-06; First posted 2012-11-14 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Exposure to Secondhand Smoke in Neonatal Infants
Keywords: Motivational Incentives; Motivational Interviewing; Secondhand Smoke; Neonatal Intensive Care Unit; NICU; High respiratory risk infants; Low birth weight infants; Environmental Tobacco Smoke; Smoking; Contingency management; Infants; Children
MeSH Terms: conditions — Smoking | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational Interviewing plus Incentives (Experimental)
  Interventions: Behavioral: Motivational Interviewing plus Incentives
- Conventional Care (CC) (Other)
  Interventions: Behavioral: Conventional Care (CC)

INTERVENTIONS:
Behavioral: Motivational Interviewing plus Incentives — 1. Two hospital-based, face-to-face MI+ sessions
  2. Two home-based MI+ sessions
  3. Attendance at each session and for the establishment of a household smoking ban at two timepoints post-discharge
  Arms: Motivational Interviewing plus Incentives
Behavioral: Conventional Care (CC) — Participants in this arm will receive brochures and a brief information meeting in the NICU.
  Arms: Conventional Care (CC)

SUMMARY:
A randomized, controlled, parallel group design will be used to test whether a Secondhand Smoke Exposure program initiated in the hospital and completed in the home using motivational interviewing plus motivational incentives (MI+) is more effective than Conventional Care (CC) with Neonatal Incentives Care Unit Infants' parents.

ELIGIBILITY:
Inclusion Criteria:

* Have an infant that is at least 1 week prior to the estimated date of hospital discharge in the NICU at Children's Memorial Hermann Hospital (CMHH)
* Report at least one person living in the home who smokes
* Agree to attend intervention sessions and to invite other household members
* Live within 50 miles of our center
* Have access to a telephone.

Exclusion Criteria:

* Severe cognitive, and/or psychiatric impairment, per judgment of NICU and research staff, that precludes cooperation with study protocol
* Inability to read, write, and speak English or Spanish
* Inability or unwillingness to provide signed consent for participation
* Inability or unwillingness to meet study requirements, including home visits for data collection and intervention purposes.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Infant Second-Hand Smoke Exposure via Urine Cotinine | Follow-up visit 4 months post-treatment
  Infant Second-Hand Smoke Exposure (SHSe) measures will be determined via urine cotinine.

SECONDARY OUTCOMES:
Secondhand Smoke Exposure outcomes | Change from Baseline to the 4 months post-treatment followup
  Primary caregiver reports via the Timeline Follow-Back and household air nicotine monitors. Number of cigarettes smoked outdoors vs. indoor and the implementation of household smoking bans will also be assessed. Primary caregivers will complete the SHSe related interviews and self-report questionnaires. Primary caregivers who are smokers will complete measures related to smoking and smoking cessation.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Stotts, PhD, Principal Investigator — University of Texas at Houston Family and Community Medicine
Locations (1):
- Children's Memorial Hermann Hospital, Houston, Texas, United States

REFERENCES:
- [Derived] Stotts AL, Northrup TF, Green C, Suchting R, Hovell MF, Khan A, Villarreal YR, Schmitz JM, Velasquez MM, Hammond SK, Hoh E, Tyson J. Reducing Tobacco Smoke Exposure in High-Risk Infants: A Randomized, Controlled Trial. J Pediatr. 2020 Mar;218:35-41.e1. doi: 10.1016/j.jpeds.2019.10.070. Epub 2019 Dec 20. PMID 31870605